CLINICAL TRIAL: NCT05369091
Title: Salivary Bmp-2 Levels And Radiographic Measurement Of Bone Density At Extracted Tooth Socket In Patients With And Without Topical Application Of Simvastatin
Brief Title: Salivary Bmp-2 Levels & Radiographic Measurement Of Bone Density at Extracted Tooth
Acronym: salivaryBMP2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Postgraduate Medical Institute, Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Mutahir Mehdi, M.Phil Oral Biology Trainee, Postgraduate Medical Institute, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M.Phil Oral Biology Trainee
Record Dates: First submitted 2022-03-29; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Bone Injury
Keywords: Simvastatin; Salivary BMP-2; Radiographic Bone density
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (No Intervention): Atraumatic Extraction Only (placement of gelatin sponge mixed with normal saline without SIMVASTATIN).
- Simvastatin (Experimental): Atraumatic Extraction and administration of SIMVASTATIN (10 mg tablet grounded and added with normal saline, with gelatin sponge as a transporter) into the socket.
  Interventions: Drug: Simvastatin 10mg

INTERVENTIONS:
Drug: Simvastatin 10mg — Atraumatic Extraction and administration of SIM (10 mg tablet grounded and added with normal saline, with gelatin sponge as a transporter) into the socket to observe alveolar bone healing.
  Other Names: SIM
  Arms: Simvastatin

SUMMARY:
Salivary Bmp-2 Levels & Radiographic Measurement Of Bone Density were evaluated At Extracted Tooth Socket in patients With & Without topical Application Of Simvastatin

DETAILED DESCRIPTION:
Objective: The objective of this study was to compare:

'The salivary BMP-2 levels in the experimental and the control groups with and without topical simvastatin application on wound of extracted tooth socket.

The bone density at extracted tooth socket by measuring mean gray value from Intra oral periapical (IOPA) radiographs in the experimental and the control groups.

Method: Twenty four patients either male or female without any systemic disease, aged between 18 years to 25 years were selected. The patients were equally divided by random computer generated numbers into experimental and control groups. In the experimental group, tooth extraction was followed by placement of simvastatin (containing 10 mg of drug). In the control group, only tooth extraction was done. Saliva sample was collected from patients on days 0, 3, 7 and 40 and levels of salivary biomarker BMP-2 were measured with the ELISA technique. IOPA radiographs were taken on days 0 and 40 to determine the bone density by measuring mean gray values with the help of ImageJ software. The data was entered in SPSS version 25 and analyzed. P-value of ≤ 0.05 was considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients with permanent dentition, age (18 years to 25 years) were considered.
* Patients undergoing extraction of maxillary or mandibular Pre molars for orthodontic procedure.
* Teeth which required only simple non surgical extraction only under local anesthesia.

Exclusion Criteria:

* Subjects taking antibiotics or non-steroidal anti inflammatory drugs (NSAIDS) within one week.
* Patients with oral mucosal lesions (leukoplakia, erythroplakia, lichen planus).
* Patients with oral carcinoma.
* Patients with xerostomia.
* Previous history of radiotherapy or chemotherapy
* Patient with known hypersensitivity to anti inflammatory drugs.
* Diabetic patients.
* Pregnant and lactating patients.
* Patients with social habits such as cigarette smoking and alcohol consumption.
* Teeth radiographically involved in any abscess/cyst/granuloma.
* Teeth requiring open surgical transalveolar extraction.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-10-03 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Salivary BMP-2 Levels | At start of study
  Mean values were measured using ELISA technique
Salivary BMP-2 Levels | At 3rd day Of Study
  Mean values were measured using ELISA technique
Salivary BMP-2 Levels | At 10th Day of study
  Mean values were measured using ELISA technique
Salivary BMP-2 Levels | At 40th Day of study
  Mean values were measured using ELISA technique
Bone Density | At start of study
  Mean grey value were measured using imageJ software
Bone Density | At 40th day of study
  Mean grey value were measured using imageJ software

CONTACTS AND LOCATIONS:
Overall Officials: shagufta nasreen, Study Chair — Pgmi. Lahore
Locations (1):
- Dental Department of Lahore General Hospital., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided